CLINICAL TRIAL: NCT00156455
Title: Sleep Disordered Breathing in Children With Single Ventricle Physiology
Status: Withdrawn | Type: Observational
Why Stopped: lack of study personel
Sponsor: University of Rochester (Other)
Responsible Party: Margaret-Ann Carno, PhD RN, University of Rochester
Other Study IDs: 10185
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Hypoplastic Left Heart Syndrome; Obstructive Sleep Apnea Syndrome; Single Ventricle Physiology
Keywords: Children; Hypoplastic left heart syndrome; Obstructive Sleep Apnea Syndrome; Single Ventricle Physiology
MeSH Terms: conditions — Hypoplastic Left Heart Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an exploratory study designed to evaluate the incidence of, and to quantify sleep disordered breathing following stage I Norwood reconstructive surgery. Sleep disordered breathing will be correlated with:

1. Elevations in pulmonary vasculature resistance at the time of Stage II surgery.
2. Risks of death

DETAILED DESCRIPTION:
This is an exploratory study designed to evaluate the incidence of, and to quantify sleep disordered breathing following stage I Norwood reconstructive surgery. Sleep disordered breathing will be correlated with:

1. Elevations in pulmonary vasculature resistance at the time of Stage II surgery.
2. Risks of death

Children with single ventricle physiology are exquisitely sensitive to alterations in pulmonary vascular resistance. Following their first operative repair (stage I Norwood), performed in their first week of life, pulmonary and systemic circulations are in parallel rather than series. As such, elevations in pulmonary vascular resistance can result in severe arterial desaturation. Additionally, elevated pre-operative pulmonary artery pressure is directly correlated with poor survival following the third and final operative repair (stage III Norwood, or Fontan).

Periodic breathing is a normal breathing pattern in sleeping infants. At the other end of the spectrum is sleep apnea. In between lies a continuum of sleep disordered breathing. Obstructive sleep apnea has an incidence of approximately 2% in children, and is associated with pulmonary and systemic hypertension. Specific studies of the incidence and effects of sleep disordered breathing in congenital heart disease are lacking. Otherwise normal children have baseline oxygen saturation in the high 90's, thereby placing them on the flat part of the oxyhemoglobin curve. But children with cyanotic congenital heart disease live with baseline oxygen saturations in the mid 70's, so that they exist on the steep part of the oxyhemoglobin dissociation curve. We hypothesize therefore that these patients are at increased risk for the hemodynamic variations occurring during apneas/hypopneas even when they are more subtle, namely during sleep disordered breathing.

We hypothesize that children who have completed stage I Norwood will experience more significant arterial desaturations during sleep associated apneic events (due to the concurrent elevation in pulmonary arterial pressure) than their normal counterparts. Additionally we hypothesize that children who experience more frequent apneic events during sleep will have elevated pre-operative pulmonary artery pressures and therefore worse outcome following stage II Norwood. Thus, we speculate that children who have completed stage I Norwood are more prone to the risks of sleep disordered breathing.

Autonomic regulation, mediated in part by aortic arch baroreceptors, is undoubtedly disrupted by the extensive surgical reconstruction required at the aortic arch during stage I Norwood palliation. Adults and children with severe sleep disordered breathing (obstructive sleep apnea) have impaired cardiac autonomic control, and increased cardiac electrical instability, with greater occurrence of ventricular arrhythmias. Apneic events place a hypoxic, mechanical and adrenergic load on the cardiovascular system thereby directly resulting in ventricular dysrhythmias. Observed late deaths following stage I Norwood are usually postulated to be secondary to fatal arrhythmias. Thus, we hypothesize that children who experience more frequent apneic events during sleep will have an increased risk of interstage mortality.

Sleep disordered breathing is a readily treatable condition in the pediatric population. Non-invasive, continuous positive airway pressure applied via a nasal mask is effective in treating sleep disordered breathing in infants. Thus, if sleep disordered breathing is identified, effective treatment is available and may reduce the risk of inter-stage mortality and adverse hemodynamics in this medically fragile population.

ELIGIBILITY:
Inclusion Criteria:

* Infants with single ventricle physiology Parents who can read and write English

Exclusion Criteria:

* Infants who are not medically stable Parents who cannot read and write English

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with hypoplasic heart condition
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-09; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi V. Connolly, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States